CLINICAL TRIAL: NCT03860090
Title: Prospective Randomized Comparison of Efficacy and Safety in Pacemaker and Defibrillator Implantation Via Cephalic Versus Axillary Vein Access. The CEPHAX Study.
Brief Title: Efficacy and Safety in Pacemaker and Defibrillator Implantation Via Cephalic Versus Axillary Vein Access (CEPHAX)
Acronym: CEPHAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A-276
Record Dates: First submitted 2019-02-21; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Pacemakers; Defibrillators; Complication; Pacemaker Electrode Lead Fracture
Keywords: Cephalic Vein; Axillary Vein
MeSH Terms: interventions — Defibrillators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AXILLARY VEIN ACCESS (Active Comparator): This group of subjects will receive the implant of device via fluoroscopy-guided axillary puncture technique.
  Interventions: Device: Pacemaker implant; Device: Defibrillator implant; Procedure: AXILLARY VEIN ACCESS
- CEPHALIC VEIN ACCESS (Active Comparator): This group of subjects will receive the implant of device via optimized cephalic vein cutdown technique.
  Interventions: Device: Pacemaker implant; Device: Defibrillator implant; Procedure: CEPHALIC VEIN ACCESS

INTERVENTIONS:
Device: Pacemaker implant — Implantation of endovenous cardiac stimulation device.
Device: Defibrillator implant — Implantation of endovenous cardiac defibrillation device.
Procedure: AXILLARY VEIN ACCESS — Fluoroscopy-guided axillary puncture to get vein access
  Arms: AXILLARY VEIN ACCESS
Procedure: CEPHALIC VEIN ACCESS — Optimized cephalic vein cutdown to get vein access
  Arms: CEPHALIC VEIN ACCESS

SUMMARY:
This clinical trial evaluates the efficacy and safety of axillary versus cephalic venous access in the pacemakers and defibrillators implantation.

Half of participants will receive the implant via fluoroscopy guided axillary venous access and the other half will receive the implant via improved cephalic venous access.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a endovenous pacemaker or defibrillator indication.

Exclusion Criteria:

* Pre-existing ipsilateral pacing electrode.
* Previous ipsilateral lymphadenectomy.
* Indication of cardiac resynchronization therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Implant Success | 30 days
  Success of the implant through the assigned access vein
Implant Complications | 30 days
  All implant related complications

SECONDARY OUTCOMES:
Lead Complications | From date of implant until the date of first documented, assessed up to 48 months
  Lead fracture or dysfunction
Upper limb thrombosis | From date of implant until the date of first documented, assessed up to 48 months
  Thrombosis of the ipsilateral upper limb
Pneumothorax | 30 days
  Implant related pneumothorax
Bleeding | 30 days
  Implant related bleeding

OTHER OUTCOMES:
Time to access. | From cutaneous incision to reach the right atrium with the guidewire, assessed up to 45 minutes.
  Time until reaching venous access.
Time of implant. | From the skin incision to the skin suture, assessed up to 180 minutes.
  Intervention time.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Jiménez Díaz, Dr., Principal Investigator — Arrhythmia Unit Director
Locations (1):
- Hospital General Universitario de Ciudad Real, Ciudad Real, Spain

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] Calkins H, Ramza BM, Brinker J, Atiga W, Donahue K, Nsah E, Taylor E, Halperin H, Lawrence JH, Tomaselli G, Berger RD. Prospective randomized comparison of the safety and effectiveness of placement of endocardial pacemaker and defibrillator leads using the extrathoracic subclavian vein guided by contrast venography versus the cephalic approach. Pacing Clin Electrophysiol. 2001 Apr;24(4 Pt 1):456-64. doi: 10.1046/j.1460-9592.2001.00456.x. PMID 11341082
- [Background] Squara F, Tomi J, Scarlatti D, Theodore G, Moceri P, Ferrari E. Self-taught axillary vein access without venography for pacemaker implantation: prospective randomized comparison with the cephalic vein access. Europace. 2017 Dec 1;19(12):2001-2006. doi: 10.1093/europace/euw363. PMID 28064251
- [Derived] Jimenez-Diaz J, Higuera-Sobrino F, Piqueras-Flores J, Perez-Diaz P, Gonzalez-Marin MA. Fluoroscopy-guided axillary vein access vs cephalic vein access in pacemaker and defibrillator implantation: Randomized clinical trial of efficacy and safety. J Cardiovasc Electrophysiol. 2019 Sep;30(9):1588-1593. doi: 10.1111/jce.14060. Epub 2019 Jul 23. PMID 31310038

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03860090/Prot_SAP_000.pdf